CLINICAL TRIAL: NCT07092800
Title: Care Pathways and Disparities in Care for Older Patients With Cancer: Typology, Determinants and Effect on Prognosis ( PASSAGE )
Acronym: PASSAGE
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Inria, the French National Institute for computer science and applied mathematics (Unknown); CentraleSupelec School of Engineering (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP240996; CSE-24-08_PASSAGE (Other: Institutional Review Board (IRB) of the AP-HP's Clinical Data Warehouse (CDW))
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Tumor; Health Services Research; Causality; Geriatric Assessment; Aged; Cancer
Keywords: Frailty; care pathways; cancer; ageing
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 70 or over with solid cancer: The following inclusion criteria will be applied to identify the study population:
  * Patients aged 70 or over,
  * Having at least one International Classification of Disease, 10th revision (ICD-10) code for solid cancer recorded as principal diagnostic or related,
  * During treatment in an AP-HP hospital,
  * Between 01/08/2017 and 31/07/2023.

SUMMARY:
More than half of new cases of cancer in Europe in 2022 occurred in people aged over 70. In addition to cancer, the majority of older people have one or more illnesses that may interact with the treatment decision, cancer progression, tolerance and efficacy of treatments, quality of life, care pathway and survival. Furthermore, cancer treatments are most often evaluated in middle-aged subjects without severe disease, so the real-life management of older patients is often empirical.

The general objective of the PASSAGE project is to assess the hospital care pathways of older patients with cancer treated at AP-HP by evaluating key elements of these pathways from both geriatric and therapeutic perspectives. Characterizing these care trajectories will help identify the most vulnerable patient profiles and potential disparities in access to care, with the goal of optimizing the management of elderly patients with cancer.

The aims of this research are 1) to provide a better description of trends in the management of older cancer patients in routine clinical practice, and 2) to assess the impact of frailty, multimorbidity and the management of these patients on the prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 or over,
* Having at least one International Classification of Disease, 10th revision (ICD-10) for solid cancer recorded as principal diagnostic or related,
* During treatment in an AP-HP hospital,
* Between 01/08/2017 and 31/07/2023.

Exclusion Criteria:

* opposition to the reuse of healthcare data

Ages: 70 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly cancer patients treated at AP-HP
Sampling Method: Probability Sample
Enrollment: 75000 (Estimated)
Dates: Start 2024-09-07 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
type of care pathway | from cancer diagnosis during a year of follow-up
  The primary endpoint is the type of care pathway as identified by longitudinal clustering analysis of Electronic Health Record (EHR) data in the year following diagnosis (medical diagnoses, procedures, admissions, treatment received),.

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor Hospital, Créteil, VAL DE Marne, France

IPD SHARING:
Plan to Share IPD: No
Data are available upon reasonable request. Proposals should be directed to ASSISTANCE PUBLIQUE HOPITAUX DE PARIS (AP-HP), Department for Clinical Research, Innovation (DRCI) represented by Mr Milan LAZAREVIC , Director. To gain access, data requestors will need to sign a data transfert agreement with the sponsor